CLINICAL TRIAL: NCT06156865
Title: Neuroimaging Reveals Treatment-related Changes in DLD: A Randomized Controlled Trial (Supplement)
Brief Title: Using Neuroimaging and Behavioral Assessments to Understand Late Talking
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Toronto (Other)
Collaborators: Holland Bloorview Kids Rehabilitation Hospital (Other); Children's Hospital Medical Center, Cincinnati (Other); University of Cincinnati (Other); Georgetown University (Other)
Responsible Party: Principal Investigator, Karla Washington, Associate Professor, University of Toronto
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 3R01DC019337-04S1 (NIH)
Record Dates: First submitted 2023-11-10; First posted 2023-12-05 (Actual); Last update posted 2025-05-11 (Actual); Status verified 2025-05

CONDITIONS: Developmental Language Disorder; Language Delay; Language Development
Keywords: children; late talking; typical development; assessment; intervention; neuroimaging
MeSH Terms: conditions — Language Development Disorders

STUDY DESIGN:
Intervention Model Description: toddlers who are late talking receive either intervention or are waitlist controls. There is also a group of typically developing children
Who Masked: Outcomes Assessor
Masking Description: the scorers of the outcomes are not informed of participants' group status
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention to address late talking (Experimental): half the participants receive an intervention program addressing late talking. The intervention is comprised of adult learning (to teach parents) and direct support for children who are late talkers. The intervention occurs over 6 to 8 weeks and is designed to improve grammar, vocabulary, and functional communication
  Interventions: Behavioral: Intervention to address late talking
- Waitlist controls (No Intervention): half the participants are waitlist controls who receive intervention at a later date, after the study has ended

INTERVENTIONS:
Behavioral: Intervention to address late talking — this intervention is designed to support both speech and language development in children who are toddlers. Given the age group of children their parents are part of the intervention program. Importantly the frequency of the intervention can range from once to twice per week, with timing also designed to complement the particular agency
  Arms: Intervention to address late talking

SUMMARY:
Late talkers (LT), representing 10-20% of children under 3, demonstrate hallmark syntax and vocabulary deficits similar to preschoolers with developmental language disorder. While effective and early interventions can mitigate the impact of late talking, not enough is known about its neural basis, yet is needed to inform the design of more individualized interventions. This proposed effort uses neuroimaging, along with behavioral methods, with the goal of better understanding the memory-language mechanisms that underlie learning and late talking, while also considering their association to treatment-related changes in LT.

DETAILED DESCRIPTION:
Late talking represents one of the most common reasons children under 3-years of age are referred for speech-language evaluations, impacting about 10%-20% of children in this age-group. Late talkers (LT) also share similarities with children diagnosed with developmental language disorder (DLD) at 4 - 5 years of age, endorsing the notion that shared neurobiological underpinnings might exist between these two clinical groups. However, little is known about the neural basis of late talking, yet is needed to better inform the design of efficacious therapies that address hallmark delays in syntax and vocabulary. For the DLD population, domain-general processes relating memory and language are being investigated in the parent grant, offering valuable testing ground for also advancing the current knowledge base regarding LT. The Procedural circuit Deficit Hypothesis (PDH) posits that relative strengths and weaknesses exist between procedural (impaired) and declarative (less impaired) memory systems. Structural abnormalities in connections between frontal brain regions and basal ganglia, with under activation and reduced connectivity also evident. However, cortical and subcortical regions in the temporal lobes, including hippocampus, might be impaired to a lesser degree.

This proposed research will use diffusion imaging to describe the neural basis (structural connectivity) of late talking and treatment-related change by way of the PDH. The investigators will gather data regarding LT before, after, and following a break in standard intervention for LT (e.g., parent coaching, direct therapy for children who are LT): LT treatment. The investigators will also include a "business as usual": LT no treatment as part of a highly feasible pragmatic design that leverages existing pipelines. The investigators will also include typically developing (TD) peers to inform development vs late talking. The central hypothesis is that treatment designed to improve syntax and vocabulary will change procedural and declarative networks in association with increases in language function and the degree of improvement may be associated with the underlying neurobiology of baseline syntax and vocabulary deficits.

Building on a robust history of recruitment and treatment of toddlers by the investigators' partnering sites, and the investigators' successful imaging partner, this project will enroll 30 LT (n=15 treatment; n=15 controls) and 15 TD peers. Aim 1 will establish the structural connectivity in LT and their TD peers between regions in the procedural learning and declarative networks. In Aim 2, the investigators will establish the neurobiological basis of treatment-related changes in LT only. The investigators examine potential changes in structural connectivity between regions of the procedural learning and declarative memory networks, and investigate whether treatment-related changes occur into the typical range (LT, TD). To meet the scientific goals, the investigators pair behavioral tools (syntax and vocabulary) with neuroimaging to describe co-occurring behavioral performance underlying learning and outcome, while also gathering parental and clinician qualitative data regarding treatment outcomes. This research will contribute novel insights into mechanisms underlying learning and impairment to offer a ground-breaking shift in the understanding of LT.

ELIGIBILITY:
Inclusion Criteria:

* child and parent are monolingual/native (primarily) English speakers
* child is enrolled at one of the participating facilities
* child is recruited via word of mouth, including social media
* child is between 18 and 30 months of age
* child does not have any contraindications to magnetic resonance imaging (i.e., intracranial metal implants, claustrophobia)
* child does not have any uncorrected vision challenges

Exclusion Criteria:

* Child does not meet criteria for LT or typical development
* Standard magnetic resonance imaging exclusion criteria
* Gestational age less than 37 weeks or greater than 42 weeks
* Special education placement of child based on ability or behavior

Ages: 18 Months to 30 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 45 (Estimated)
Dates: Start 2024-01-19 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Aim 1/Pre - Structural connectivity data using diffusion imaging | Weeks 1 to 2 (Time 1/pre)
  Connectivity data (density of streamlines connecting regions of the procedural learning and declarative networks) will be measured using tractography, a 3D modeling technique, to visually represent nerve tracts using data that we collect using diffusion MRI from each of the 45 participants at Weeks 1 to 2 as part of a non-sedated sleep scan.
Aim 2/Pre - Changes in structural connectivity data using diffusion imaging | Weeks 1 to 8 or 9 (pre to post); Weeks 10 to 17 or 18 (post to followup)
  Changes in connectivity data (density of streamlines connecting regions of the procedural learning and declarative networks) calculated using data collected over two time points (pre to post; post to followup) will be measured from each of the 45 participants. Connectivity data measured using tractography collected using diffusion MRI are gathered from these participants at pre, post, and followup to inform these changes over time as part of a non-sedated sleep scan.

SECONDARY OUTCOMES:
Aim 1/Pre - Raw score on the MacArthur Bates Communicative Development Inventories: Words and Sentences- (first set) | Weeks 1 to 2 (Time 1/pre - first set)
  Raw score data calculated using the MacArthur Bates Communicative Development Inventories: Words and Sentences. This measure is completed by each of the 45 children's parents. High scores indicate better performance compared to lower scores. Minimum score is '0' and maximum is '680'. These data serve as main secondary outcomes.
Aim 1 - Raw score on the Focus on the Outcomes of Communication Under Six Parent Version- (second set) | Weeks 1 to 2 - (Time 1/pre - second set)
  Raw score data calculated using the Focus on the Outcomes of Communication Under - Parent Version. This measure is completed by each of the 45 children's parents. High scores indicate better performance compared to lower scores. Minimum score is '0' and maximum is '238'. These data will inform main secondary outcomes.
Aim 1/Pre - Raw score on the Focus on the Outcomes of Communication Under Six Clinician Version- (third set) | Weeks 1 to 2 - (Time 1/pre - third set)
  Raw score data calculated using the Focus on the Outcomes of Communication Under - Clinician Version. This measure is completed by each of the 45 children's clinicians. High scores indicate better performance compared to lower scores. Minimum score is '0' and maximum is '238'. These data will inform main secondary outcomes.
Aim 1/Pre - Raw score on the Intelligibility in Context Scale- (fourth set) | Weeks 1 to 2 - (Time 1/pre - fourth set)
  Raw score data calculated using the Intelligibility in Context Scale. This measure is completed by each of the 45 children's parents. High scores indicate better performance compared to lower scores. Minimum score is '0' and maximum is '35'. These data will inform additional secondary outcomes.
Aim 1/Pre - Raw score on the Communication Function Classification System- (fifth set) | Weeks 1 to 2 - (Time 1/pre - fifth set)
  Raw score data obtained using the Communication Function Classification System. This measure is completed by each of the 45 children's parents. Lower scores indicate better performance compared to higher scores. The minimum score is "1" and the maximum is "5". These data will inform additional secondary outcomes.
Aim 1/Pre - Raw score calculated using a Consonant Inventory- (sixth set) | Weeks 1 to 2 - (Time 1/pre - sixth set)
  Raw score data obtained using a Consonant Inventory collected during a play-based language sample. These data are collected from each of the 45 children during their assessment with the clinician. Higher scores indicate better performance compared to lower scores. The minimum score is "0" and the maximum score is "24". These data will inform additional secondary outcomes.
Aim 1/Pre - Raw score calculated using a Play-based language sample- (seventh set) | Weeks 1 to 2 - (Time 1/pre - seventh set)
  Raw score data obtained on language complexity (grammar and vocabulary) collected during a play-based language sample timed for 15-minutes. These data are collected from each of the 45 children during their assessment with the clinician. Higher scores indicate better performance compared to lower scores. The minimum score is "0" and the maximum score is variable. There is not a ceiling since this is based on a spontaneous language sample and some children can talk more than others during the 15-minute period. However we have a metric of performance based on scores less than the 10th percentile and then those greater than the 10th percentile. Performance at or below the 10th percentile is worse than performance greater than the 10th percentile. These data will inform additional secondary outcomes.
Aim 2 - Changes in structural connectivity data using diffusion imaging for late talkers only | Weeks 1 to 8 or 9 (pre to post); Weeks 10 to 17 or 18 (post to followup)
  Changes in connectivity data (density of streamlines connecting regions of the procedural learning and declarative networks) calculated using data collected over two time points (pre to post; post to followup) will be measured from only the 30 participants who are late talkers. Connectivity data measured using tractography collected using diffusion MRI are gathered from these participants at pre, post, and followup to inform these changes over time as part of a non-sedated sleep scan.
Aim 2 - Raw score changes on the MacArthur Bates Communicative Development Inventories: Words and Sentences- (first set) | Weeks 1 to 8 or 9 (pre to post); Weeks 10 to 17 or 18 (post to followup)
  Raw change score data calculated using the MacArthur Bates Communicative Development Inventories: Words and Sentences that is completed at pre, post, followup. This measure is completed on three occasions by the 30 parents whose children are late talkers. High change scores indicate better performance compared to lower change scores. The minimum score is "0" and the maximum score is "680". These data serve as main secondary outcomes to inform immediate (pre-post) and maintenance of changes (post-followup).
Aim 2 - Raw score changes on the Focus on the Outcomes of Communication Under Six Parent Version- (second set) | Weeks 1 to 8 or 9 (pre to post); Weeks 10 to 17 or 18 (post to followup)
  Raw change score data calculated using the Focus on the Outcomes of Communication Under Six that is completed at pre, post, followup. This measure is completed on three occasions by the 30 parents whose children are late talkers. High change scores indicate better performance compared to lower change scores. The minimum score is "0" and the maximum score is "238". These data serve as main secondary outcomes to inform immediate (pre-post) and maintenance of changes (post-followup).
Aim 2 - Raw score changes on the Focus on the Outcomes of Communication Under Six Clinician Version- (third set) | Weeks 1 to 8 or 9 (pre to post); Weeks 10 to 17 or 18 (post to followup)
  Raw change score data calculated using the Focus on the Outcomes of Communication Under Six that is completed at pre, post, followup. This measure is completed on three occasions by the clinicians of the 30 children who are late talkers. High change scores indicate better performance compared to lower change scores. The minimum score is "0" and the maximum score is "238". These data serve as main secondary outcomes to inform immediate (pre-post) and maintenance of changes (post-followup).
Aim 2 - Raw score changes on the Intelligibility in Context Scale- (fourth set) | Weeks 1 to 8 or 9 (pre to post); Weeks 10 to 17 or 18 (post to followup)
  Raw change score data calculated using the Intelligibility in Context Scale that is completed at pre, post, followup. This measure is completed on three occasions by the 30 parents whose children are late talkers. High change scores indicate better performance compared to lower change scores. The minimum score is "0" and the maximum score is "35". These data serve as additional secondary outcomes to inform immediate (pre-post) and maintenance of changes (post-followup).
Aim 2 - Raw score changes on the Communication Function Classification System- CFCS (fifth set) | Weeks 1 to 8 or 9 (pre to post); Weeks 10 to 17 or 18 (post to followup)
  Raw change score data calculated using the Communication Function Classification System that is completed at pre, post, followup. This measure is completed on three occasions by the 30 parents whose children are late talkers. Higher change scores indicate better performance compared to lower change scores. The minimum score is "1" and the maximum score is "5". These data serve as additional secondary outcomes to inform immediate (pre-post) and maintenance of changes (post-followup).
Aim 2 - Raw score changes in the Consonant Inventory- (sixth set) | Weeks 1 to 8 or 9 (pre to post); Weeks 10 to 17 or 18 (post to followup)
  Raw change score data obtained using a Consonant Inventory collected during a play-based language sample that is completed at pre, post, followup. These data are collected on three occasions from the 30 children who are late talkers. Higher change scores indicate better performance compared to lower change scores. The minimum score is "0" and the maximum score is "24". These data serve as additional secondary outcomes to inform immediate (pre-post) and maintenance of changes (post-followup).
Aim 2 - Raw change scores calculated using a Play-based language sample- (seventh set) | Weeks 1 to 8 or 9 (pre to post); Weeks 10 to 17 or 18 (post to followup)
  Raw change score data obtained on language complexity (grammar and vocabulary). These data are calculated during a play-based language sample that is completed with a clinician at pre, post, followup. These data are collected on three occasions from the 30 children who are late talkers. Higher change scores indicate better performance compared to lower change scores. The minimum score is "0" and the maximum score is variable. There is not a ceiling since this is based on a spontaneous language sample and some children can talk more than others during the 15-minute period. However we have a metric of performance based on scores less than the 10th percentile and then those greater than the 10th percentile. Performance at or below the 10th percentile is worse than performance greater than the 10th percentile. These data serve as additional secondary outcomes to inform immediate (pre-post) and maintenance of changes (post-followup).
Aim 2 - Raw change scores calculated using the MacArthur Bates Communicative Development Inventories- (eighth set) | Weeks 1 to 8 or 9 (pre to post); Weeks 10 to 17 or 18 (post to followup)
  Raw change score data calculated using the MacArthur Bates Communicative Development Inventories: Words and Sentences that is completed at pre, post, followup. This measure is completed on three occasions by the 30 parents of children who are late talkers as well as by the 15 parents of typically developing peers. High change scores indicate better performance compared to lower change scores. The minimum score is "0" and the maximum score is "680". These data serve as additional secondary outcomes to inform immediate (pre-post) and maintenance of changes (post-followup).
Raw change scores calculated using the Focus on the Outcomes of Communication Under Six Parent Version- (ninth set) | Weeks 1 to 8 or 9 (pre to post); Weeks 10 to 17 or 18 (post to followup)
  Raw change score data calculated using the Focus on the Outcomes of Communication Under Six Parent Version that is completed at pre, post, followup. This measure is completed on three occasions by the 30 parents of children who are late talkers as well as by the 15 parents of typically developing peers. High change scores indicate better performance compared to lower change scores. The minimum score is "0" and the maximum score is "238". These data serve as additional secondary outcomes to inform immediate (pre-post) and maintenance of changes (post-followup).
Raw change scores calculated using the Focus on the Outcomes of Communication Under Six Clinician Version- (tenth set) | Weeks 1 to 8 or 9 (pre to post); Weeks 10 to 17 or 18 (post to followup)
  Raw change score data calculated using the Focus on the Outcomes of Communication Under Six Clinician Version that is completed at pre, post, followup. This measure is completed on three occasions by the clinicians of 30 children who are late talkers as well as by clinicians of 15 typically developing peers. High change scores indicate better performance compared to lower change scores. The minimum score is "0" and the maximum score is "238". These data serve as additional secondary outcomes to inform immediate (pre-post) and maintenance of changes (post-followup).

OTHER OUTCOMES:
Aim 1/Pre - qualitative data clinician reported | Weeks 1 to 2 (Pre/Time 1)
  Other outcomes using themes from qualitative questions to the clinicians of the 45 participants. Scores on a scale are not used in this qualitative effort.
Aim 1/Pre - qualitative data parent reported | Weeks 1 to 2 (Pre/Time 1)
  Other outcomes using themes from qualitative questions to the parents of each of the 45 participants. Scores on a scale are not used in this qualitative effort.
Aim 2 - Qualitative data parent reported | Weeks 1 or 2 (pre/Time 1); Weeks 9 or 10 (post/Time 2), Weeks 17 or 18 (followup/Time 3)
  Other outcomes using themes from qualitative questions to the parents of each of the 30 children who are late talkers. These qualitative data are collected at three time points: pre, post, followup. Scores on a scale are not used in this qualitative effort.
Aim 2 - qualitative data clinician reported | Weeks 1 or 2 (pre/Time 1); Weeks 9 or 10 (post/Time 2), Weeks 17 or 18 (followup/Time 3)
  Other outcomes using themes from qualitative questions to the clinicians of the 30 children who are late talkers. These qualitative data are collected at three time points: pre, post, followup. Scores on a scale are not used in this qualitative effort.

CONTACTS AND LOCATIONS:
Overall Officials: Karla N Washington, PhD, Principal Investigator — University of Toronto
Locations (2):
- Canada (2):
  - Grandview Kids, Oshawa, Ontario
  - Speech Specialists, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: Yes
The proposed research will include a sample of late talkers (LT), typically developing (TD) peers, and their parents recruited through the community programs in Ontario Canada. The dataset will include paper-based data along with neuroimaging data, in accordance with Research Ethics Board approval, including parent consent regarding the sharing of data. Further, data are expected to be video- and audio-recorded for reliability and data analyses. While the final dataset will be de-identified, we believe that the possibility of identification remains due to the use of video- and audio- recorded aspects of this research. Thus, we will only make the paper-based and neuroimaging data available only under a data-sharing agreement, which applies a higher-level of permission (parent-approved), with the provisos in place
Supporting Information: Analytic Code
Time Frame: In keeping with our Resource Sharing Plan with the NIH, we agree to make data available is specific repositories 12 to 24-months after the end of the research project timeline associated with the supplement award mechanism
Access Criteria: We intend to share data with researchers, clinicians, and government/educational officials, including at academic institutions. These individuals will work with institutions/entities that have necessary Ethics Boards and Federal Wide Assurance. We agree to institute an adjudication process for granting or denying access to data that includes procedures consistent with the NIH data sharing policies. Requesting individuals will be asked to provide a request in writing that adheres to set components. They will be able to access the data for educational (student training) and research (secondary analyses) purposes regarding intervention outcomes and syntax and vocabulary language-learning profiles in LT and TD peers. We agree that the names of individuals and their institutions/entities will be summarized in the annual report regardless of whether or not these persons are granted or denied permission to access the data.